CLINICAL TRIAL: NCT05547022
Title: Critical Limb Ischemia in Trinidad and Tobago- A Series of 157 Endovascular Limb Salvage Attempts in Patients With CLTI
Brief Title: Endovascular Limb Salvage in Trinidad and Tobago
Status: Completed | Type: Observational
Sponsor: Naveen Seecheran (Other)
Responsible Party: Sponsor-Investigator, Naveen Seecheran, Senior Lecturer, The University of The West Indies
Organization: The University of The West Indies (Other)
Other Study IDs: CEC175/04/17
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Limb Salvage Rates With Endovascular Therapy
Keywords: Critical limb-threatening ischemia (CLTI); Endovascular revascularization (EVR); Peripheral arterial disease (PAD); Peripheral vascular disease (PVD).
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critical Limb ischemia patients with tissue loss: CLI patients with minor and major tissue loss who had endovascular revascularisation
  Interventions: Procedure: Endovascular revascularisation

INTERVENTIONS:
Procedure: Endovascular revascularisation — Peripheral vascular angioplasty or stenting

SUMMARY:
The purpose of this study was to investigate limb salvage rates in patients with critical limb ischemia after endovascular revascularization.

DETAILED DESCRIPTION:
A retrospective analytical study assessing limb salvage attempts and outcomes in 157 consecutive patients with CLI and tissue loss. It was for the period of May 2018 and May 2021 at Eric Williams Medical Sciences Complex.

The objectives of this study include Primary: To determine the success rate of target lesion revascularisation using endovascular limb salvage techniques in Critical limb ischemia patients with minor and major tissue loss.

Secondary objectives included:

1. to compare and contrast limb salvage rate to international standards
2. to assess the maintenance of amputation-free survival and bipedal ambulation
3. to evaluate the angiosome concept and its effect on wound healing
4. to evaluate primary patency rate
5. to assess the overall morbidity and mortality of endovascular treatment for critical limb ischemia
6. to observe the outcomes of various wound healing techniques and its efficacy

ELIGIBILITY:
Inclusion Criteria:

CLI patient with tissue loss who underwent infra inguinal endovascular limb salvage

Exclusion Criteria:

CLI patients with tissue loss who had surgical bypass CLI patients with no tissue loss

Ages: 33 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are recruited from EWMSC, Trinidad who presented with CLI.
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Primary outcome | 2 to 3 years
  to determine the success rate of target lesion revascularization using endovascular limb salvage techniques

OTHER OUTCOMES:
Secondary Outcome | 2 to 3 years
  to assess the maintenance of amputation free survival and bipedal ambulation
Co-Secondary Outcome | 2 to 3 years
  to evaluate primary patency rate

CONTACTS AND LOCATIONS:
Locations (1):
- Eric Williams Medical Sciences Complex, Port of Spain, North Central, Trinidad and Tobago

REFERENCES:
- [Derived] Harnanan D, Parbhu S, Pran L, Baboolal I, Harnarayan P, Naraynsingh V, Seecheran N. Endovascular Revascularization and Outcomes of Critical Limb-Threatening Ischemia in Trinidad and Tobago: The EVENT Pilot Study-Challenges in a Limited-Resource, Caribbean Setting. Cardiol Ther. 2023 Sep;12(3):511-524. doi: 10.1007/s40119-023-00322-9. Epub 2023 Jun 17. PMID 37329412